CLINICAL TRIAL: NCT06581744
Title: Non Invasive Imaging Methods for Detecting Primary Aldosteronism： a Clinical Positron EmissionTomography (PET) Study of 18F-Pentixather
Brief Title: Non Invasive Imaging Methods for Detecting PA：a Clinical PET Study of 18F-Pentixather
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fangfang Sun (Other)
Responsible Party: Sponsor-Investigator, Fangfang Sun, Pharmacist, The First Affiliated Hospital of Dalian Medical University
Organization: The First Affiliated Hospital of Dalian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYX001
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: Primary aldosteronism; Radiation Dosimetry; 18F-Pentixather
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hyperaldosteronism (Experimental): Intravenous inject 18F-Pentixather，perform PET/CT imaging at the designated time
  Interventions: Other: [18F]AlF-NOTA-Pentixather

INTERVENTIONS:
Other: [18F]AlF-NOTA-Pentixather — inject 185~370MBq [18F]AlF-NOTA-Pentixather

SUMMARY:
Primary aldosteronism (PA) is the most common endocrine cause of hypertension. 68Ga-pentixafor PET/CT possesses a relatively high sensitivity and specificity for Aldosterone producing adenoma (APA) detection. However, 68Ga is usually eluted from a 68Ge-68Ga generator, only a small amount of isotopes can be achieved once time. [18F]AlF-chelation is a promising strategy that would solve these issues. 18F labeled Pentixafor-Based Imaging Agent([18F]AlF-NOTA-Pentixather) has been reported by Andreas Poschenrieder. [18F]AlF-NOTA-Pentixather displayed high and CXCR4-specific in vivo uptake in Daudi xenografts (13.9%±0.8% injected dose per gram [ID/g] at 1 hour post injection[p.i.]). But to date 18F-Pentixather has not been studied in humans. In this program the investigators will estimate the radiation dosimetry of [18F]AlF-NOTA-Pentixather, evaluate the sensitivity and specificity of the [18F]AlF-NOTA-Pentixather as a probe for APA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with primary aldosteronism and willing to undergo surgery
2. Clinically highly suspected of primary aldosteronism, but the diagnostic test cannot clearly identify the patients
3. Postoperative recurrence in patients with primary aldosteronism

Exclusion Criteria:

1. Pregnant and lactating women.
2. Patients with poor autonomous behavior ability, severe claustrophobia, and critically ill patients requiring life support who are unable to cooperate in completing the examination.
3. There are other situations where patients are not suitable for this examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of radiation dosimetry and biodistribution of 18F-Pentixather determined with PET/CT in Patients with PA | 6 month
  Images were acquired using a Biograph Truepoint 64 PET/CT scanner (Siemens, Erlangen, Germany).The dosimetry analysis was performed using 3d-slicer（version 5.6.1, with slicerOpenDose3D module (https://gitlab.com/opendose/opendose3d). OpenDose: open access resources for nuclear medicine dosimetry (www.opendose.org).
Analyze the specificity and sensitivity of 18F-pentixather PET/CT for the diagnosis of APA | 3 years
  Compare the 18F-Pentixather SUVmax with the CXCR4，CYP11B2 immunohistochemical score. Calculate the sensitivity and specificity of 18F-pentixafor PET/CT results for an indication of APA, IAH, or NFA lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng Y, Long T, Peng N, Zhen M, Ye Q, Zhang Z, He Y, Chen Z, Gan Y, Luo M, Li C, Liu Z, Guo M, Wang M, Luo X, Hu S, Liu L, Jiang T. The Value of Targeting CXCR4 With 68Ga-Pentixafor PET/CT for Subtyping Primary Aldosteronism. J Clin Endocrinol Metab. 2023 Dec 21;109(1):171-182. doi: 10.1210/clinem/dgad421. PMID 37477496
- [Result] Gao Y, Ding J, Cui Y, Li T, Sun H, Zhao D, Zhang Y, Huo L, Tong A. Functional nodules in primary aldosteronism: identification of CXCR4 expression with 68Ga-pentixafor PET/CT. Eur Radiol. 2023 Feb;33(2):996-1003. doi: 10.1007/s00330-022-09058-x. Epub 2022 Sep 7. PMID 36070092